CLINICAL TRIAL: NCT05803174
Title: Screening and Identification of Biomarkers for High Myopia by a Rapid Method
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Beijing Tongren Hospital (Other)
Collaborators: Tsinghua University (Other)
Responsible Party: Sponsor
Other Study IDs: 010133
Record Dates: First submitted 2023-03-26; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: High Myopia
Keywords: biomarkers
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Emmetropic subjects: Spherical equivalent (Diopter, D) to be between -0.5 and +0.5 D
  Interventions: Diagnostic Test: blood sample
- Low and moderate myopic subjects: Spherical equivalent (Diopter, D) to be less than -0.5 but over -6.0D
  Interventions: Diagnostic Test: blood sample
- High myopic subjects: Spherical equivalent (Diopter, D) to be over or equal to -6.0D
  Interventions: Diagnostic Test: blood sample

INTERVENTIONS:
Diagnostic Test: blood sample — Blood collection Circulating serum concentrations of melatonin and dopamine were determined from fasting blood samples. Participants were required to fast from 10 pm the previous evening. A 5 mL serum blood sample was collected from the antecubital vein between 8.30 am and 10 am.
  Tear collection Tear samples were collected using Schirmer's strip without anesthesia between 8:30-10:00am. Tears were extracted in 200 μl of 1 X Phosphate Buffered Saline with 0.1% Tween-20 (PBST).
  Saliva collection Saliva samples were collected via the "passive drool" method with subjects in a seated position. Subjects were asked to rinse their mouth with water 10 minutes prior to saliva collection and to refrain from using lip makeup during the sampling period.
  Other Names: saliva, tear fluid

SUMMARY:
To screen and identify sensitive biomarkers for high myopia via a robust, convenient, and cost-effective approach according to the association between high myopia and concentration of biomarkers in tear fluid, saliva and blood among adults and children.

DETAILED DESCRIPTION:
Myopia has emerged as a serious public health issue, with the prevalence increasing rapidly worldwide, especially in East Asia. Increasingly early onset of myopia leads to high myopia with sight-threatening complications (e.g., secondary cataracts, glaucoma, and retinal detachment) that cannot be treated by optical means.

A key goal of myopia research over the past decades has been to identify those sensitive biomarkers. Accurate monitoring of myopic-specific biomarkers is desirable for achieving early diagnosis, progression assessment, and prognostic management.

However, measurement of levels of MMPs in human have been restricted to aqueous humors, which is invasive and the findings are difficult to be replicated in other studies. In order to achieve the goal of convenient high myopic detection, the use of a panel of biomarkers using a multiplex approach may indeed be rapid and highly reproducible with potentially higher sensitivity and specificity than single biomarkers, such as MMP 2 for the early detection of high myopia.

In this study we have used a newly developed immunoassay technology, and identified a panel of novel biomarkers for early detection of high myopia by non-invasively evaluating several biomarkers that are measurable in the saliva and tear fluid of adults.

ELIGIBILITY:
Children Inclusion Criteria

1. Children aged 6-17
2. Removing flexible lenses for at least 1 week, flexible astigmatism and hard lenses for at least 3 weeks, orthokeratology lenses for at least 3 months;
3. Best corrected visual acuity of either eye were all ≥ 1.0;
4. The range of myopia in either eye was -15 D ≤ SE ≤ +1.0 D;
5. Astigmatism of either eye less than -5.0 D;
6. Anisometropia ≤ -1.5 D;
7. There was no active ocular inflammatory diseases; no obvious corneal cloud or macula, anormal corneal topography, and no tendency of keratoconus.
8. Intraocular pressure of either eye is of 10 to 21 mmHg;
9. On the basis of full understanding, children and their guardians sign the informed consent;

Adults Inclusion Criteria

1. adults aged 18-35
2. Removing flexible lenses for at least 1 week, flexible astigmatism and hard lenses for at least 3 weeks, orthokeratology lenses for at least 3 months;
3. Best corrected visual acuity of either eye were all ≥ 1.0;
4. The range of myopia in either eye was -15 D ≤ SE ≤ +1.0 D;
5. Astigmatism of either eye less than -5.0 D;
6. Anisometropia ≤ -1.5 D;
7. There was no active ocular inflammatory diseases; no obvious corneal cloud or macula, anormal corneal topography, and no tendency of keratoconus.
8. Intraocular pressure of either eye is of 10 to 21 mmHg;
9. On the basis of full understanding, adults sign the informed consent;

Exclusion Criteria:

1. Amblyopia: best corrected visual acuity (BCVA) of either eye less than 1.0 for adults and children over 6 years old;
2. Active ocular inflammatory diseases, such as uveitis and other inflammatory diseases;
3. Secondary myopia, genetic disease or connective tissue- related myopia;
4. Moderate or severe ptosis;
5. Congenital cataract, glaucoma;
6. Other fundus diseases other than myopic related fundus lesions;
7. Intraocular or refractive surgery history;
8. The refractive medium is turbid, and it is impossible to take a clear fundus image; (9)Unable to cooperate with fundus image shooting and other examination;

(10)Do not receive cycloplegia or have contraindications; (11)Poor overall condition, unable to follow up for a long time; (12)The subject refuses to participate in the research; (13)Other cases in which the researcher judges that it is not suitable for participation in the study.

Ages: 6 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: There are two levels of research, namely children and adults. Each level is divided into three groups of 20 subjects each. So about 120 subjects are anticipated in total. Taken into account the proportion of exclusion, 150 subjects are invited to recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of TNF-α in tear fluid, saliva and blood sample among emmetropic, low and moderate myopic, and high myopic groups | June 30, 2023
  TNF-α: Tumor necrosis factor is an adipokine and a cytokine.

SECONDARY OUTCOMES:
Concentration of IL-1 in tear fluid, saliva and blood sample among emmetropic, low and moderate myopic, and high myopic groups | June 30, 2023
  IL-1: Interleukin 1

OTHER OUTCOMES:
Concentration of IL-10 in tear fluid, saliva and blood sample among emmetropic, low and moderate myopic, and high myopic groups | June 30, 2023
  IL-10: Interleukin 10, an anti-inflammatory cytokine
Concentration of IL-6 in tear fluid, saliva and blood sample among emmetropic, low and moderate myopic, and high myopic groups | June 30, 2023
  IL-6: Interleukin 6, a pro-inflammatory cytokine
Concentration of TIMP in tear fluid, saliva and blood sample among emmetropic, low and moderate myopic, and high myopic groups | June 30, 2023
  TIMP: Tissue inhibitor of metalloproteinases, a family of proteins that act as enzyme inhibitors
Concentration of MMP2 in tear fluid, saliva and blood sample among emmetropic, low and moderate myopic, and high myopic groups | June 30, 2023
  MMP2: Proteins of the matrix metalloproteinase (MMP) family are involved in the breakdown of extracellular matrix in normal physiological processes
Concentration of EGF in tear fluid, saliva and blood sample among emmetropic, low and moderate myopic, and high myopic groups | June 30, 2023
  EGF:Epidermal growth factor (EGF) is a protein that stimulates cell growth.

CONTACTS AND LOCATIONS:
Overall Officials: Shi-Ming Li, Principal Investigator — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No